CLINICAL TRIAL: NCT01569230
Title: Clinical Trial to Evaluate and Compare the Efficacy and Safety of Individualized and Standardized Acupuncture for Knee Osteoarthritis Patients: Randomized, Single-blind, Controlled Study
Brief Title: Efficacy and Safety Study of Individualized and Standardized Acupuncture Treatment for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eun Jung Kim (Other)
Collaborators: Semyung University (Other); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Eun Jung Kim, Research professor, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B080017-KCT0000385
Record Dates: First submitted 2012-03-26; First posted 2012-04-03 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis Knee
Keywords: Knee osteoarthritis; acupuncture; sham acupuncture
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Individualized acupuncture (Experimental): The patients in this group received individualized acupuncture prescribed by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 2 years of clinical experience. The acupuncture formulas were composed based on the pattern diagnosis, which is an unique diagnosis system of Oriental Medicine.
  Interventions: Procedure: Individualized Acupuncture
- Standardized Acupuncture (Experimental): The patients in this group received standardized acupuncture treatment using the same acupuncture points, applied by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 2 years of clinical experience. The acupuncture formulas were composed based on literature review of RCTs.
  Interventions: Procedure: Standardized Acupuncture
- Sham acupuncture (Sham Comparator): Non-penetrating acupuncture device, Park-sham acupuncture, was applied to the patients. The appearance of the acupuncture is same but the needles do not penetrate the skin.
  Interventions: Procedure: sham acupuncture
- Waiting (No Intervention): No interventions were applied to the patients in this group. Only assessments were made at each visit.
  Interventions: Other: Waiting

INTERVENTIONS:
Procedure: Standardized Acupuncture — The treatment was applied twice a week for 20 minutes for 6 weeks(12sessions) 9 Acupuncture points(SP9,GB34, ST36, ST35, Xiyan(EX-LE5), BL60, GB39, SP6 and KI3)were used for all the patients assigned to this group. Sterile Stainless Steel(25mm x 40mm) disposable acupuncture needles manufactured by Dong-Bang Acupuncture Co.(Korea) were used.
  Arms: Standardized Acupuncture
Procedure: sham acupuncture — The treatment was applied twice a week for 6 weeks(12sessions). The sham acupuncture was applied on the 9 same acupuncture points as in the standardized acupuncture group. Each session was 20 minutes long
  Other Names: Park Sham Device
  Arms: Sham acupuncture
Procedure: Individualized Acupuncture — The treatment was applied twice a week for 20 minutes for 6 weeks(12sessions)
  Arms: Individualized acupuncture
Other: Waiting — No interventions were applied to the patients in this group.
  Other Names: No interventions
  Arms: Waiting

SUMMARY:
The purpose of this study is to verify the efficacy and safety of acupuncture treatments (Individualized, Standardized acupuncture) for patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
The investigators targeted the patients with knee OA. After treatment in 4 groups - individualized acupuncture treatment, standardized acupuncture treatment, sham-needle treatment, and waiting groups - the investigators will compare the effects of pain relieving and daily performing improvement. So the investigators will confirm the efficacy of acupuncture, and further the best treatment method. In addition, the investigators are going to evaluate the safety of abnormal reaction during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age, but below 80 years of age
2. Knee pain from OA in one or both knees in the last 3 months or more
3. Presence of knee OA diagnosed by an orthopedist based on American College of Rheumatology classification criteria
4. Knee pain from OA in one or both knees rated > 4 cm on a 10 cm Visual Analog Scale (VAS)
5. An understanding of the objectives and methods of the clinical trial, and willingness in completing the consent form.
6. Those who are reliable and willing to cooperate in this test, and obey the restrictions for the next 3 months

Exclusion Criteria:

1. Trauma to or surgery on the knee(s) within 6 months prior to enrollment, causing pain or functional problems
2. A history of prolotherapy, injection of hyaluronic acid or cortisone within the last 3 months
3. A physical or laboratory finding indicating infection, presence of an autoimmune disease, or inflammatory arthritis
4. Serious organic disease, and severe dysfunction due to the medical illness (e.g. Arrhythmia, Angina pectoris, Stroke, Asthma, etc.)
5. More severe pain in regions other than the knee joint.
6. Pregnant
7. When researchers evaluate that it is not appropriate to participate in this clinical test

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities) Scale change | at 2nd(Baseline),8(after 3weeks of treatment),13th(after 6 weeks of treatment) and 14(follow up evaluation after 6 weeks from the last treatment) visit
  WOMAC scale is checked by the patients. WOMAC scale is a tool to check of the disability, stiffness and pain by knee pain.

SECONDARY OUTCOMES:
100mm Pain Visual Analogue Scale | at 2(Baseline), 3, 4, 5, 6, 7, 8(after 3weeks of treatment), 9, 10, 11, 12, 13(after 6 weeks of treatment), and 14th(follow up evaluation after 6 weeks from the last treatment) visit
  The patient is asked to indicate their perceived pain intensity along a 100 mm horizontal line, where '0' represents 'no pain' and '100', 'unbearable pain'.
6 Minute walk test | at 2nd(Baseline),8(after 3weeks of treatment),13th(after 6 weeks of treatment) and 14(follow up evaluation after 6 weeks from the last treatment) visit
  the distance of subject's 6 Minute walking
WOMAC pain | at 2(Baseline), 3, 4, 5, 6, 7, 8(after 3weeks of treatment), 9, 10, 11, 12, 13(after 6 weeks of treatment), and 14th(follow up evaluation after 6 weeks from the last treatment) visit
  The pain part of WOMAC (Westren Ontario and McMaster Universities) Scale
Investigator global assessment(IGA) | at 2(Baseline), 3, 4, 5, 6, 7, 8(after 3weeks of treatment), 9, 10, 11, 12, 13(after 6 weeks of treatment), and 14th(follow up evaluation after 6 weeks from the last treatment) visit
  5 Grading of Investigator(1=Very good, 2=good, 3=fair, 4=poor, 5=very poor)
Patient global assessment(PGA) | at 2(Baseline), 3, 4, 5, 6, 7, 8(after 3weeks of treatment), 9, 10, 11, 12, 13(after 6 weeks of treatment), and 14th(follow up evaluation after 6 weeks from the last treatment) visit
  5 Grading of Investigator(1=Very good, 2=good, 3=fair, 4=poor, 5=very poor)
Adverse Events | at 2(Baseline), 3, 4, 5, 6, 7, 8(after 3weeks of treatment), 9, 10, 11, 12, 13th(end of treatment) visit
  Any unpredicted symptoms were checked at each follow up visit and if any, the symptom, time of occurrence, and length of duration were recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kap-Sung Kim, Ph.D., Principal Investigator — Donnguk University Oriental Medical center
Locations (1):
- Donnguk University Oriental Medical center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim EJ, Lim CY, Lee EY, Lee SD, Kim KS. Comparing the effects of individualized, standard, sham and no acupuncture in the treatment of knee osteoarthritis: a multicenter randomized controlled trial. Trials. 2013 May 7;14:129. doi: 10.1186/1745-6215-14-129. PMID 23782709